CLINICAL TRIAL: NCT07183956
Title: Comparison of the Silverman-Andersen Score and the Downes Score in Assessing the Severity of Respiratory Distress and Predicting Noninvasive Ventilation Failure in Neonates
Brief Title: Comparison of the Silverman-Andersen Score and the Downes Score
Acronym: CSASDS
Status: Not yet recruiting | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ozkan Ilhan, Associate Professor, Muğla Sıtkı Koçman University
Other Study IDs: MSKU-NICU-OI-02
Record Dates: First submitted 2025-09-06; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Distress Neonatal; Noninvasive Ventilation; Intubation; Scoring Systems
Keywords: Silverman-Andersen score; Downes score; Newborn; Respiratory distress; Noninvasive ventilation
MeSH Terms: conditions — Hyaline Membrane Disease; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants >28 weeks GA treated with NIPPV due to respiratory distress within the first 12 h of life: Infants born at >28 weeks of gestation who develop respiratory distress within the first 6 h of life and receive noninvasive ventilation therapy (NIPPV) within the first 12 h will be included in the study. Silverman-Andersen and Downes scores will be assessed 20-30 minutes after initiation of NIPPV using standardized scoring systems. Blood gas analysis will be performed within 30 minutes after NIPPV initiation. Additional indices of respiratory severity-including the respiratory severity score (RSS), FiO₂, mean airway pressure (MAP), and oxygen saturation index (OSI)-will be recorded at 20-30 minutes. RSS will be calculated as FiO₂ × MAP; MAP as [(Ti × PIP) + (Te × PEEP)] / (Ti + Te); and OSI as [MAP (cmH₂O) × FiO₂ (%)] / SpO₂ (%)] (18, 19). NIPPV failure will be defined as the need for intubation in an infant receiving NIPPV. In the same infants, the predictive value of the Silverman-Andersen score and the Downes score for NIPPV failure at 24 hours and 72 hours will be evaluated.

SUMMARY:
This study aimed to compare the Silverman-Andersen score and the Downes score in predicting noninvasive ventilation (NIPPV) failure in preterm and term infants who received NIPPV support due to postnatal respiratory distress, as well as to evaluate the agreement of these scoring systems with other methods used to assess the severity of respiratory distress.

The present study was designed as a prospective, multicenter, observational study conducted with neonates undergoing noninvasive ventilation.

DETAILED DESCRIPTION:
The present study was designed as a prospective, multicenter, observational study conducted with neonates undergoing noninvasive ventilation. The study will be conducted in 4 centers (Mugla Training and Research Hospital, Mugla, Turkey; Akdeniz University School of Medicine, Antalya, Turkey; Antalya Training and Research Hospital, Antalya, Turkey; Sanliurfa Training and Research Hospital, Sanliurfa, Turkey). Written informed consent will be obtained from the parents of each neonatal patient prior to enrollment in the study.

Participants:

Preterm infants born at >28 weeks of gestation and term infants born at ≥37 weeks of gestation who developed respiratory distress within the first 6 hours after birth (defined as the presence of at least two of the following: respiratory rate ≥60/min, subcostal/intercostal retractions, and grunting), whose respiratory distress persisted for more than 6 hours, who were within the first 12 hours of life, had a Silverman-Andersen score ≥3, and received NIPPV support will be included in the study (1).

Infants with major congenital malformations, airway or pulmonary anomalies, cardiovascular or respiratory instability due to sepsis, cyanotic congenital heart disease, severe intraventricular hemorrhage, contraindications for NIPPV therapy (such as congenital nasal anomalies, congenital diaphragmatic hernia, or abdominal wall defects), those who required intubation or chest compressions in the delivery room, required intubation within the first hour of life, died within the first 24 hours of life, were born at ≤28 weeks of gestation, or were diagnosed with air leak syndrome (pneumothorax) prior to initiation of NIPPV therapy will be excluded from the study.

Respiratory support protocol Infants ≥34 weeks of gestation with respiratory distress within the first 6 hours of life will be observed for 2 hours; if distress persists and the Silverman-Andersen score is ≥3, NIPPV will be initiated. Infants <34 weeks with respiratory distress and a Silverman-Andersen score ≥3 will be directly started on NIPPV. NIPPV is a routine, noninvasive respiratory support modality widely used in our unit and globally. Ventilatory support will be delivered via short binasal prongs using a mechanical ventilator.

Initial NIPPV settings will be: PIP 15-20 cmH₂O, PEEP 5-6 cmH₂O, rate 40-50 breaths/min, inspiratory time (Ti) 0.35-0.45 s, and flow 8-10 L/min. PIP may be increased by 1-2 cmH₂O increments up to a maximum of 25 cmH₂O if required. FiO₂ will be titrated to maintain oxygen saturation between 90-94%.

Assessment of respiratory severity Silverman-Andersen and Downes scores will be assessed 20-30 minutes after initiation of NIPPV using standardized scoring systems. Blood gas analysis will be performed within 30 minutes after NIPPV initiation. Additional indices of respiratory severity-including the respiratory severity score (RSS), FiO₂, mean airway pressure (MAP), and oxygen saturation index (OSI)-will be recorded at 20-30 minutes. RSS will be calculated as FiO₂ × MAP; MAP as [(Ti × PIP) + (Te × PEEP)] / (Ti + Te); and OSI as [MAP (cmH₂O) × FiO₂ (%)] / SpO₂ (%)] (18, 19). All scoring and calculations will be performed by a pediatrician, neonatology fellow, or neonatologist, each trained in standardized assessment prior to the study.

Definition of NIPPV failure and success NIPPV failure will be defined as the presence of severe respiratory acidosis (pH <7.20, PaCO₂ >60 mmHg), oxygen saturation <90% despite FiO₂ >50%, >3 apnea episodes within 1 hour, >2 apnea episodes requiring positive pressure ventilation with a bag-valve-mask device within 24 hours, or shock requiring inotropic support. Infants with NIPPV failure will be intubated and managed with conventional mechanical ventilation. Infants extubated within 1 hour following ENSURE (ENtubation, SURfactant, Extubation) will not be considered NIPPV failures, whereas those remaining intubated for >1 hour after ENSURE will be classified as failures.

Weaning from NIPPV will be attempted when PIP is reduced to 14-15 cmH₂O, PEEP to 5 cmH₂O, respiratory rate to 20-30/min, and FiO₂ <30%, provided that the Silverman-Andersen score is <3 and both clinical findings and blood gas parameters are acceptable. Infants successfully weaned from NIPPV will be considered to have achieved NIPPV success.

Surfactant and caffeine therapy Surfactant therapy is routinely performed in our unit and is not a novel intervention. Surfactant will be administered at a dose of 200 mg/kg via either LISA (Less Invasive Surfactant Administration) or ENSURE when FiO₂ ≥40% is required to maintain target oxygen saturation of 90-94%. In preterm infants with RDS who require intubation for respiratory failure, surfactant will be administered via an endotracheal tube (2). A second dose will be given if FiO₂ requirement persists at ≥40%. All infants born before 32 weeks of gestation or with a birth weight <1500 g will routinely receive prophylactic caffeine therapy as standard practice.

Study parameters and outcomes The following parameters will be compared between infants with and without NIPPV failure: Silverman-Andersen score, Downes score, respiratory severity score, oxygen saturation index, SpO₂/FiO₂ ratio, duration of NIPPV, surfactant requirement, mortality, blood gas parameters, and demographic characteristics.

The primary outcome is to determine the most appropriate scoring system for predicting noninvasive ventilation failure by comparing the predictive performance of the Silverman-Andersen and Downes scores within the first 24 and 72 hours of life. The secondary outcome is to assess the correlation of both scores with duration of noninvasive ventilation, SpO₂/FiO₂ ratio, oxygen saturation index, respiratory severity score, and blood gas parameters (pH and PaCO₂), and to determine which scoring system demonstrates stronger correlation. Additionally, the predictive value of both scores for mortality and surfactant requirement in infants born before 34 weeks of gestation will be compared.

Sample size calculation Previous studies have shown that initiating respiratory support with NIPPV in infants with respiratory distress reduces the incidence of respiratory failure and the need for intubation compared to NCPAP (3). Permatahati et al. (4) reported an NCPAP failure rate of 37% when applied as primary respiratory support in preterm infants with respiratory distress. In the present study, the investigators hypothesized that the NIPPV failure rate would decrease from 37% to 20% when NIPPV is used as the primary respiratory support in neonates with respiratory distress. Based on this hypothesis, a power analysis was performed using G*Power version 3.1.9.4, with a type I error of 5% and 80% power, resulting in a required sample size of 220 patients.

Statistical analysis:

Data will be analyzed using the SPSS statistical software. Descriptive statistics will be presented as percentages (%), means, or medians, as appropriate. The Kolmogorov-Smirnov, Shapiro-Wilk, skewness, and kurtosis tests will be used to assess the normality of the data. Comparisons between infants with and without NIPPV failure will be performed using the Student's t-test, Mann-Whitney U test, and chi-square test, as appropriate.

Receiver operating characteristic (ROC) curve analysis will be used to calculate the area under the curve (AUC), sensitivity, and specificity of the Silverman-Andersen and Downes scores for predicting NIPPV failure. Comparisons of AUC values will be performed using MedCalc software. Optimal cut-off values for both scores in predicting NIPPV failure will be determined using the maximum Youden index.

Pearson and Spearman correlation analyses will be used to assess the relationship between the Silverman-Andersen and Downes scores and other respiratory distress parameters, including respiratory severity score, oxygen saturation index, blood gas pH and PaCO₂, and SpO₂/FiO₂ ratio. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at >28 weeks of gestation or term infants born at ≥37 weeks of gestation.
* Development of respiratory distress within the first 6 hours after birth, defined as the presence of at least two of the following: Respiratory rate ≥60/min, Subcostal/intercostal retractions, Grunting.
* Persistence of respiratory distress for more than 6 hours.
* Age within the first 12 hours of life.
* Silverman-Andersen score ≥3.
* Receiving NIPPV support.

Exclusion Criteria:

* Major congenital malformations.
* Airway or pulmonary anomalies.
* Cardiovascular or respiratory instability due to sepsis.
* Cyanotic congenital heart disease.
* Severe intraventricular hemorrhage.
* Contraindications for NIPPV therapy (e.g., congenital nasal anomalies, congenital diaphragmatic hernia, abdominal wall defects).
* Requirement of intubation or chest compressions in the delivery room.
* Requirement of intubation within the first hour of life.
* Death within the first 24 hours of life.
* Gestational age ≤28 weeks.
* Diagnosis of air leak syndrome (pneumothorax) prior to initiation of NIPPV therapy.

Ages: 2 Hours to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born at >28 weeks of gestation and term infants born at ≥37 weeks of gestation who developed respiratory distress within the first 6 hours after birth.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
To determine the predictive role of the Silverman-Andersen score for noninvasive ventilation failure at 24 and 72 hours of life. | 24 hours and 72 hours after birth
  Noninvasive ventilation failure will be defined as the need for intubation in an infant receiving NIPPV. The Silverman-Andersen score will be assessed at 30 minutes after initiation of NIPPV therapy, and its predictive value for noninvasive ventilation failure will be evaluated at 24 and 72 hours of life. The Silverman-Andersen score assesses upper chest movement, intercostal retractions, subxiphoid retractions, nasal flaring, and air entry to the lungs on auscultation. Each parameter is scored between 0 and 2, yielding a total score ranging from 0 to 10. Higher scores indicate greater severity of respiratory distress (5).
To determine the predictive role of the Downes score for noninvasive ventilation failure at 24 and 72 hours of life | 24 hours and 72 hours after birth
  Noninvasive ventilation failure will be defined as the need for intubation in an infant receiving NIPPV. The Downes score will be assessed at 30 minutes after initiation of NIPPV therapy, and its predictive value for noninvasive ventilation failure will be evaluated at 24 and 72 hours of life. The Downes score evaluates cyanosis, respiratory rate, retractions, grunting, and air entry to the lungs on auscultation. Each parameter is scored between 0 and 2, yielding a total score ranging from 0 to 10. Higher scores indicate greater severity of respiratory distress (5).

SECONDARY OUTCOMES:
Agreement of the Respiratory Severity Score with the Silverman-Andersen score and Downes score | 30 minutes after the initiation of NIPPV therapy
  Respiratory Severity Score will be calculated as FiO₂ × MAP (mean airway pressure) (references: 6, 7).
Agreement of the oxygen saturation index (OSI) with the Silverman-Andersen score and Downes score | 30 minutes after the initiation of NIPPV therapy
  Oxygen saturation index (OSI) will be calculated following formula: [MAP (cmH₂O) × FiO₂ (%)] / SpO₂ (%)] (references: 6, 7).
Agreement of the blood gas pH and PaCO₂ with the Silverman-Andersen score and Downes score | 30 minutes after the initiation of NIPPV therapy
  The investigators routinely perform blood gas evaluations after birth in infants with respiratory distress.
Agreement of the SpO₂/FiO₂ ratio with the Silverman-Andersen score and Downes score | 30 minutes after the initiation of NIPPV therapy
  In infants with respiratory distress, the investigators monitor SpO₂ using a bedside monitor after birth and record FiO₂ levels on the ventilator used for noninvasive ventilation follow-up
The predictive value of Silverman-Andersen score and Downes score for surfactant requirement in infants born before 34 weeks of gestation | At 48 hours following the initiation of NIPPV therapy
The predictive value of Silverman-Andersen score and Downes score for mortality , | Prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ozkan Ilhan, Study Director — Mugla Training and Research Hospital; Ozkan Ilhan, Assoc. Prof., Principal Investigator — Mugla Sitki Kocman University School of Medicine
Locations (4):
- Turkey (Türkiye) (4):
  - Akdeniz University School of Medicine, Department of Neonatology, Antalya, Antalya
  - Antalya Training and Research Hospital, Department of Neonatology, Antalya, Antalya
  - Mugla Training and Research Hospital, Department of Neonatology, Muğla, Mentese
  - Sanliurfa Training and Research Hospital, Department of Neonatology, Sanliurfa, Şanlıurfa

IPD SHARING:
Plan to Share IPD: No
Our data is available upon request, and we are committed to providing access to interested researchers for the purpose of scientific inquiry.

REFERENCES:
- [Background] Iyer NP, Mhanna MJ. Non-invasively derived respiratory severity score and oxygenation index in ventilated newborn infants. Pediatr Pulmonol. 2013 Apr;48(4):364-9. doi: 10.1002/ppul.22607. Epub 2013 Jan 28. PMID 23359457
- [Background] Muniraman HK, Song AY, Ramanathan R, Fletcher KL, Kibe R, Ding L, Lakshmanan A, Biniwale M. Evaluation of Oxygen Saturation Index Compared With Oxygenation Index in Neonates With Hypoxemic Respiratory Failure. JAMA Netw Open. 2019 Mar 1;2(3):e191179. doi: 10.1001/jamanetworkopen.2019.1179. PMID 30924897
- [Background] Abdallah Y, Mkony M, Noorani M, Moshiro R, Bakari M, Manji K. CPAP failure in the management of preterm neonates with respiratory distress syndrome where surfactant is scarce. A prospective observational study. BMC Pediatr. 2023 May 3;23(1):211. doi: 10.1186/s12887-023-04038-6. PMID 37138252
- [Background] Permatahati WI, Setyati A, Haksari EL. Predictor Factors of Continuous Positive Airway Pressure Failure in Preterm Infants with Respiratory Distress. Glob Pediatr Health. 2021 Apr 7;8:2333794X211007464. doi: 10.1177/2333794X211007464. eCollection 2021. PMID 33889679
- [Background] Lemyre B, Deguise MO, Benson P, Kirpalani H, Ekhaguere OA, Davis PG. Early nasal intermittent positive pressure ventilation (NIPPV) versus early nasal continuous positive airway pressure (NCPAP) for preterm infants. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD005384. doi: 10.1002/14651858.CD005384.pub3. PMID 37466143
- [Background] Ozkan H, Erdeve O, Kutman HGK. Turkish Neonatal Society guideline on the management of respiratory distress syndrome and surfactant treatment. Turk Pediatri Ars. 2018 Dec 25;53(Suppl 1):S45-S54. doi: 10.5152/TurkPediatriArs.2018.01806. eCollection 2018. PMID 31236018
- [Background] 1. Report of National Neonatal perinatal Database (NNPD) 2002-2003. Available from http://www.newbornwhocc.org/nnpo_html. Accessed Dec 2014.